CLINICAL TRIAL: NCT01382953
Title: The Simple ECG Monitoring Trial (Comparison of a Simple ECG Recording System With a Standard ECG Recording System for Holter Monitoring)
Brief Title: The Simple ECG Monitoring Trial (Comparison of a Novel Recording System With a Standard Holter Monitor)
Status: Completed | Type: Observational
Sponsor: Seattle Institute for Cardiac Research (Other)
Collaborators: Cardiac Science Corporation. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10131-01B
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Syncope; Pre-syncope; Atrial Fibrillation; Supraventricular Tachycardia
Keywords: Holter Monitor, Ambulatory Electrocardiography Monitoring
MeSH Terms: conditions — Syncope; Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Standard Holter/Investigational patch — The standard Holter and Investigational patch will be worn simultaneously for 24 hours. A single follow-up visit will follow in 2 days to remove both systems which will be sent away for analysis with the results of the standard system used, if pertinent, for patient management.
  Other Names: Cardiac Science Burdick Holter.; Investigational patch trilobite system.

SUMMARY:
The purpose of this research is to simplify the standard recording system of the heart rhythm. The investigators desire to improve the ease of monitoring the cardiac rhythm for 24 hours. The investigators intent is to use a very small, innovative monitoring patch system that relieves the patient of wearing a cumbersome and uncomfortable recording system. This research trial will carry the title "The Simple ECG Monitoring" for Comparison of a Sternal ECG Recording System with a Standard ECG Recording System for Holter Monitoring. The data from the investigational device is for comparative purposes only. It will not be used by medical personnel for study subject treatment or diagnostic purposes.

DETAILED DESCRIPTION:
Externally applied cardiac rhythm monitors are common tools used to diagnose symptoms that may or may not be related to cardiac rhythm abnormalities. Common problems that may lead to the use of cardiac rhythm monitors are syncope (loss of consciousness), near-syncope (near loss of consciousness), palpitations (the sensation of an abnormal heart beat), or monitoring of known cardiac rhythm problems like atrial fibrillation. The purpose of this research is to confirm the clinical value of a much easier-to-use cardiac rhythm monitoring system, hereafter referred to as the Investigational Monitoring System. Prior to discussing the investigational monitoring system, we will review standard electrocardiographic monitoring tools used to evaluate the heart's rhythm.

Excluding a routine 12 lead electrocardiogram that takes a snapshot view of the hearts electrical signal, the most common tool for monitoring the heart rhythm is a Holter monitor. A Holter monitor is also called an ambulatory cardiac monitor. A Holter monitor records every heartbeat for 24 hours. It requires wearing multiple electrodes and carrying a recording system that is usually worn on a belt or on a holster strap. Such systems are relatively bulky and difficult to conceal in public venues. Also, their electrodes often disconnect, especially during sleep when the patient is unaware of electrode detachments that can occur when turning or during exercise. Moreover, they can't be worn during showering. These shortcomings notwithstanding, standard Holters remain the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Syncope of uncertain etiology or
* Pre-syncope of uncertain etiology or
* Palpitations of uncertain etiology or
* Management of known AF/SVT patients

Exclusion Criteria:

* Any abnormal or friable skin over the anterior thorax and upper abdomen
* Sternal incision within 3 months from the date of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic referral, Cardiology Clinic, Electrophysiology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To compare the *diagnostic yield and *ECG signal quality of the standard Holter with that of the Simple ECG Monitoring patch | 24 Hours
  * Diagnostic yield is the proportion of patients for whom an arrhythmogenic source of symptoms is established, or ruled out. The two systems will be correlated following completion of blinded batch reviews.
  * ECG signal quality is scoring the ability of each system to record electrical activity from the atrium (P-waves)using the following scale: Excellent, Good, Fair, Poor, Non-existent.

SECONDARY OUTCOMES:
Skin comfort or discomfort: Was skin irritated? | 48 Hours
  User will rate skin comfort on a pre-determined scale: none, mild, moderate, severe.
  Clinician will examine and rate patient's skin irritation when device is removed, using a pre-determined scale: none, mild, moderate, severe.
Device comfort | 48 Hours
  Was device comfortable to wear? User will rate on a pre-determined scale: very uncomfortable, mildly uncomfortable, comfortable.
  Was device inconspicuous under clothing? User will rate on a pre-determined scale: conspicuous, inconspicuous.
  Was ability to sleep affected by wearing the device? User will rate on a pre-determined scale: yes, no.
Device stability and contact | 48 Hours
  Did the device stay in place in the chest location where it was attached? Clinician will evaluate visually, and rate on a pre-determined scale: yes, no.
User interface | 48 Hours
  Was the patient able to access the button on the device to 'mark' events, such as sensing an episode of palpitations? User will rate on a pre-determined scale: Yes, no.
  Did the clinician find the device easy to attach to patient? Clinician will rate on a pre-determined scale with a rating of 1 through 5: 1 = very easy to attach and 5 = very hard to attach.
  Did the clinician find the device easy to remove from the patient? Clinician will rate on a pre-determined scale with a rating of 1 through 5: 1 = very easy to remove and 5 = very hard to remove.

CONTACTS AND LOCATIONS:
Overall Officials: Gust H. Bardy, MD, Principal Investigator — Seattle Institute for Cardiac Research
Locations (4):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Gene Trobaugh Cardiology, Enumclaw, Washington
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch